CLINICAL TRIAL: NCT07380776
Title: Effects of Preoperative Education Program on Quality of Life for Patients Undergoing Cholecystectomy at Erbil Teaching Hospitals
Brief Title: Preoperative Education Program on Gastrointestinal Quality of Life in Cholecystectomy Patients
Acronym: PEP-GIQLI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, BURHAN IZZADDIN SABIR SALIH, MSc in adult Nursing (Lecturer at college of nursing / Hawler Medical University, Hawler Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GIQLI Index of cholecystectomy
Record Dates: First submitted 2026-01-24; First posted 2026-02-02 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Preoperative Patient Education , Quality of Life , Cholecystectomy
Keywords: preoperative eduaction; gallstone disease; quality of life (GIQLI)
MeSH Terms: conditions — Cholelithiasis

STUDY DESIGN:
Intervention Model Description: interventional parallel-group study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- control group (routin hospital pre operative education (Active Comparator): The routine hospital intervention provided to patients undergoing cholecystectomy is delivered by nursing staff as part of standard care. This education included a clear explanation of the indication for cholecystectomy, as well as information about the surgical procedure and type of anesthesia. Patients were instructed on pre-operative preparation, such as fasting requirements and medication management. Post-operatively, education focused on early ambulation, breathing and coughing exercises to prevent respiratory complications, and gradual resumption of physical activity.
  In addition, patients received dietary guidance emphasizing a gradual return to oral intake and the avoidance of fatty or fried foods during the recovery period. Discharge education covered medication adherence, follow-up appointments, and the importance of seeking medical attention when necessary. This routine educational intervention aimed to enhance patients' knowledge, promote recovery, and reduce postoperati
  Interventions: Other: preoperative educatinal program

INTERVENTIONS:
Other: preoperative educatinal program — The Comprehensive Pre-Operative Education program is a structured intervention designed to enhance patients' understanding of gallbladder problems and improve the quality of life of patients suffering from gallstone disease who are undergoing cholecystectomy. The program comprises two individualized education sessions lasting 45 minutes each, focusing on essential topics such as Definition of gallbladder, Main functions of the gallbladder, the common health issues that can affect the gallbladder, the types of gallstones, diagnosis of gallstones, how they are treated, and nonsurgical treatments for gallstones. Complications could potentially occur from gallbladder removal. General pre-operation patient preparation for gallbladder removal surgery, Postoperative Care After Gallbladder Removal Surgery (Cholecystectomy), Dietary Modifications After Surgery, recommendations about how to be away from aggravating factors that affect health status after surgery, discharge instructions, and ins

SUMMARY:
The goal of this clinical trial is to evaluate whether the comprehensive preoperative educational program for patients undergoing cholecystectomy can improve their knowledge and enhance postoperative quality of life compared to patients who receive routine preoperative intervention. The study focuses on patients who underwent cholecystectomy, particularly in the age range from 18 to 75 years, and aim to determine if comprehensive preoperative education has a greater impact on improving the quality of life level then routine intervention alone The main questions it aims to answer are

1. Does preoperative patient education improve postoperative quality of life scores more effectively than the routine intervention alone
2. Does the preoperative education improve the patient's knowledge and practices regarding the cholecystectomy operation? Researchers will compare patients who receive preoperative education to those receiving routine hospital intervention to assess the differences in postoperative quality of life score and patient outcomes.

Participants will:

Control group patients receive routine preoperative intervention, while the intervention group will participate in educational sessions on comprehensive preoperative education about gallstones and the cholecystectomy operation

DETAILED DESCRIPTION:
This clinical trial aims to explore the effectiveness of a preoperative health education program on knowledge and quality of life for patients undergoing cholecystectomy in surgical wards at public teaching hospitals in Erbil City, Iraq. Gallstone disease (GSD) is one of the most common leading causes of morbidity and biliary tract diseases worldwide. Gallstones constitute a significant health problem in developed societies, affecting 10% to 15% of the adult population, and are associated with a significant health and financial burden. Inadequate health education and the absence of structured preoperative counseling programs have contributed to inconsistent knowledge among patients and variable recovery outcomes following the cholecystectomy procedure.

This study will evaluate whether equipping patients who are undergoing cholecystectomy with comprehensive preoperative education enhances the postoperative quality of life and postoperative outcomes.

The study will involve two groups of patients with confirmed cholelithiasis who are undergoing cholecystectomy

Intervention group: patients receiving a comprehensive preoperative educational program will cover:

* General information about the gallbladder included nine questions covered (physiological function of GB, positive indicator signs and symptoms of gallstones, laboratory test indicators for gallstones, which gender and age groups are at higher risk of developing gallstones, common diagnostic tools, and standard methods of treatment for symptomatic patients).
* Patient information about cholecystectomy surgery included five questions covered (number of small incisions in the laparoscopic method, advantages of the laparoscopic method, absolute contraindications of cholecystectomy, situation of operation conversion from laparoscopic to open, and contraindications of both types of open and laparoscopic cholecystectomy).
* Patient's information about preoperative preparations included nine questions covering essential investigations and diagnostic tests before operation, informed consent concerning the reason for fasting before surgery, skin preparation (operative site), the appropriate type of soap for skin preparation, cosmetic use before operation, the type of medication the patients must stop before surgery, personal item removal, and the type of clothes recommended for surgery.
* Postoperative care included eight questions covered (position after surgery, postoperative complications avoided by early ambulation, gastrointestinal symptoms after surgery, normal period, can the patients return to work and daily activities, postoperative exercises such as deep breathing and coughing, leg and ankle pump exercises, ankle circle exercises, and changing position).
* Patients' information about discharge guidelines included six questions covering steps of keeping the wound area clean after surgery, the importance of avoiding soaking in pools or showers for a long time after surgery, eating times per day after surgery, nutrients recommended after surgery, signs and symptoms of wound infection, and situations that need immediate calling or visiting the physician.

The primary outcome will be the change and improvement in postoperative quality of life score and patients' outcomes over a specific period. Secondary outcomes will include patient knowledge and practice measured through a pre- and post-intervention structured questionnaire.

The participants, after one month, will attend follow-up visits where the quality of life will be assessed, and patients will be assessed for their knowledge and understanding of the preoperative educational guidance provided. Data on patients will also be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* An adult patient.
* Both genders
* Individuals' interest in participating in the study.
* Patients who were diagnosed with cholelithiasis requiring a cholecystectomy operation confirmed by ultrasound and physical examination
* Ability to attend the educational program
* Conscious patient able to communicate
* Being elective candidates for cholecystectomy

Exclusion Criteria:

* Who had participated in a previous education program regarding open and laparoscopic cholecystectomy
* Patients who refuse to complete the post-test.
* Those with professional health qualifications
* Patients with mental disabilities and mental illnesses.
* People who changed their opinion about participating in the study or missed consecutive educational intervention sessions for any reason.
* The procedure is done other than standard laparoscopic and open cholecystectomy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Improvement of the quality of life | one month (measured at baseline and at one month postoperative)
  His outcome aims to assess the differences in the level of improvement of their quality of life at the end of the intervention. The study will compare the effectiveness of a comprehensive preoperative educational program versus the routine intervention provided to patients undergoing cholecystectomy. The quality of life will be assessed by using the gastrointestinal Quality of Life Index, providing a quantitative assessment of intervention impact on postoperative quality of life

SECONDARY OUTCOMES:
improvement in the patients' knowledge about gallstone and cholecystectomy | (Before the educational intervention, and one month after the operation and education program )
  His measure will assess the change in the patient's knowledge regarding the gallstone and cholecystectomy operation before and after the education program. The assessment will be conducted using a validated structured questionnaire that gauges understanding of general information about gallbladder anatomy, cholecystectomy operation, preoperative preparation, postoperative care, and discharge guidelines after the operation.

CONTACTS AND LOCATIONS:
Locations (1):
- Hawler Medical University/College of nursing, Erbil, Kurdistan Region, Iraq

IPD SHARING:
Plan to Share IPD: No